CLINICAL TRIAL: NCT00610792
Title: An Open Label, Phase 2 Study of Biweekly VELCADE and Intermittent CAELYX in Patients With Ovarian Cancer Failing Platinum Containing Regimens
Brief Title: Phase 2 Study of Twice Weekly VELCADE and CAELYX in Patients With Ovarian Cancer Failing Platinum Containing Regimens
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never submitted to IND. Study is being sponsored by Johnson and Johnson in the EU only.
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Clinical Study Medical Monitor, Millennium Pharmaceuticals, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26866138-OVC-2001; S043VELC02
Record Dates: First submitted 2008-01-28; First posted 2008-02-08 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2009-07

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Bortezomib; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bortezomib; Drug: pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: bortezomib — 1.3 mg/m2 on Days 1, 4, 8 & 11 every 3 weeks (1 cycle = 21 days) for up to six cycles
  Other Names: VELCADE
Drug: pegylated liposomal doxorubicin — 30 mg/m2 on Day 1 every 3 weeks (1 cycle = 21 days) for up to six cycles
  Other Names: CAELYX

SUMMARY:
This a Phase 2, multicenter open label, uncontrolled 2-step design. Patients will be arranged in two groups based upon the response to their last platinum containing therapy. The two groups are, 1) Platinum Resistant Patients: patients with progressive disease while on platinum containing therapy or stable disease after at least 4 cycles; patients relapsing following an objective response while still receiving treatment; patients relapsing after an objective response within 6 months from the discontinuation of the last chemotherapy and 2) Platinum-Sensitive Patients: patients who relapsed following an objective response after 6 months from the discontinuation of platinum containing chemotherapy. All patients will receive pyridoxine at least 200mg by mouth daily beginning approximately one week prior to the initiation of the combination chemotherapy and it will continue up to the end of the last treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed diagnosis of ovarian carcinoma of epithelial origin, primary tubal or peritoneal carcinoma;
* Progressive or recurrent disease
* The following patient types based upon the disease measurability may enroll in this study and will be considered for efficacy evaluation.

Patients may have measurable disease strictly following the RECIST guidelines. CA125 levels must be obtained according to the Rustin guidelines to enable a complete evaluation of response/progressive disease according to the GCIG guidelines. Patients may enter with a solitary measurable lesion which has not been confirmed by histology/cytology. These patients will be considered evaluable for response according to a modified RECIST which will not require the histological/cytological confirmation of the lesion. CA125 levels must be obtained according to the Rustin guidelines to enable a complete evaluation of progressive disease according to the GCIG guidelines. Patients with non-measurable disease will be considered evaluable for response provided CA125 data has been collected according to the Rustin guidelines and a complete evaluation of response/progressive disease according to the GCIG guidelines maybe conducted.

* Numbers of prior chemotherapy(s): maximum 2 prior chemotherapies. Reintroduction of a platinum at relapse, after an initial response lasting > 6 months is considered 1 chemotherapy regimen only.
* ECOG performance status grade 0 or 1
* Age ≥ 18 and ≤ 75 yrs
* Adequate hematological, liver and renal function (hemoglobin ≥ 9 g/dL, absolute neutrophil count (ANC) ≥ 1.50 x 109/L; platelets ≥ 100 x 109/L, bilirubin within UNL; alkaline phosphatase ≤ 1.5 x UNL; ALT, AST ≤ UNL or ≤ 2.5 x UNL in case of liver metastases; albumin ≥ 2.5 g/dL; creatinine ≤ UNL
* Life expectancy of at least 3 months
* Prior anthracycline limited to doxorubicin equivalent of 280mg/m2 with progression free interval of at least 12 months for patients who have been pre-treated with CAELYX
* LVEF must be within normal limits
* Signed and dated informed consent

Exclusion Criteria:

* Chemotherapy, hormonal, radiation or immunotherapy or participation in any investigational drug study within 4 weeks of study entry
* Pre-existing peripheral neuropathy > Grade 1
* Presence of cirrhosis or active or chronic hepatitis
* Presence of serious cardiac (congestive heart failure, angina pectoris, myocardial infarction within one year prior to study entry, uncontrolled hypertension or arrhythmia), neurological or psychiatric disorder
* Presence of uncontrolled intercurrent illness or any condition which in the judgment of the Investigator would place the subject at undue risk or interfere with the results of the study
* Symptomatic brain metastases or leptomeningeal disease
* Pregnancy or lactation or unwillingness to use adequate method of birth control
* Active infection
* Known history of allergy to mannitol, boron or liposomally formulated drugs.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Estimated)
Dates: Start 2006-07; Primary Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
tumor response, as measured using the Gynecologic Cancer Intergroup (GCIG) recommendations (modified RECIST); duration of response and progression free interval | baseline scans performed up to 4 weeks prior to start of treatment; further assessments at end of cycle 2; confirmation is required

SECONDARY OUTCOMES:
Overall safety profile of the combination characterized by type, frequency, severity, timing and relationship to study therapy of adverse events and laboratory abnormalities (NCI-CTCAE V3.0) | Patients followed for adverse events for 30 days after the last drug administration, or until all drug related toxicities and ongoing SAEs havebeen resolved

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (7):
- Italy (4):
  - Division of Gynecologic Oncology, Università Catholica Sacre Cuore, Campbasso
  - Istituto Europeo di Oncologia (IEO), Milan
  - Istituto Nazionale dei Tumori, Milan
  - Dept. Procreational Medicine, Università di Pisa, Pisa
- Switzerland (3):
  - Kantonsspital St. Gallen, Sankt Gallen, CH
  - Gynecologic Oncology Unit, Ospedale Sant' Anna, Turin
  - Istituto Oncologico della Svizzera Italiana, Bellinzona